CLINICAL TRIAL: NCT00552617
Title: A Multi-Center, Randomized, Open-Label, Prospective Bridging, Parallel Dose-Finding Trial Comparing Efficacy, Safety and Pharmacokinetics of 4 Doses of Org 25969 and Placebo Administered at Reappearance of T2 After Rocuronium or Vecuronium in Japanese and Caucasian Subjects. Part B: Caucasian Subjects
Brief Title: A Bridging Trial Comparing Sugammadex (Org 25969) at Reappearance of T2 in Japanese and Caucasian Participants. Part B: Caucasian Participants (P05971)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05971; 19.4.208B (Other: Organon Protocol Number); MK-8616-035 (Other: Merck Protocol Number); 2005-001133-15 (EudraCT Number)
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Rocuronium; Vecuronium Bromide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Rocuronium + Placebo (Placebo Comparator): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered intravenously (IV), followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
  Interventions: Drug: Placebo; Drug: Rocuronium
- Rocuronium + 0.5 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Rocuronium + 1.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Rocuronium + 2.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Rocuronium + 4.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Vecuronium + Placebo (Placebo Comparator): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
  Interventions: Drug: Placebo; Drug: Vecuronium
- Vecuronium + 0.5 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Vecuronium
- Vecuronium + 1.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Vecuronium
- Vecuronium + 2.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Vecuronium
- Vecuronium + 4.0 mg/kg Sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex; Drug: Vecuronium

INTERVENTIONS:
Drug: Sugammadex — After induction of anesthesia an intubation dose of (Neuromuscular blocking agent) NMBA was administered IV: either 0.9 mg/kg rocuronium or 0.1 mg/kg vecuronium.
  Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.03 mg/kg vecuronium IV could be administered if necessary.
  At reappearance of T2 the randomized single dose of sugammadex 0.5 to 4 mg/kg IV was administered
  Other Names: Org 25969
  Arms: Rocuronium + 0.5 mg/kg Sugammadex; Rocuronium + 1.0 mg/kg Sugammadex; Rocuronium + 2.0 mg/kg Sugammadex; Rocuronium + 4.0 mg/kg Sugammadex; Vecuronium + 0.5 mg/kg Sugammadex; Vecuronium + 1.0 mg/kg Sugammadex; Vecuronium + 2.0 mg/kg Sugammadex; Vecuronium + 4.0 mg/kg Sugammadex
Drug: Placebo — After induction of anesthesia an intubation dose of NMBA was administered IV: either 0.9 mg/kg rocuronium (arm 1) or 0.1 mg/kg vecuronium (arm 6).
  Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.03 mg/kg vecuronium IV could be administered if necessary.
  At reappearance of T2 the randomized single dose of Placebo IV was administered
  Arms: Rocuronium + Placebo; Vecuronium + Placebo
Drug: Rocuronium — After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV.
  Maintenance doses of 0.1-0.2 mg/kg rocuronium IV could be administered if necessary.
  Arms: Rocuronium + 0.5 mg/kg Sugammadex; Rocuronium + 1.0 mg/kg Sugammadex; Rocuronium + 2.0 mg/kg Sugammadex; Rocuronium + 4.0 mg/kg Sugammadex; Rocuronium + Placebo
Drug: Vecuronium — After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV. Maintenance doses of 0.02-0.03 mg/kg vecuronium IV could be administered if necessary.
  Arms: Vecuronium + 0.5 mg/kg Sugammadex; Vecuronium + 1.0 mg/kg Sugammadex; Vecuronium + 2.0 mg/kg Sugammadex; Vecuronium + 4.0 mg/kg Sugammadex; Vecuronium + Placebo

SUMMARY:
The objective of the trial was to establish the dose-response relation of sugammadex (Org 25969) given as a reversal agent of rocuronium or vecuronium at reappearance of T2 (the amplitude of the first response of second twitch to train of four (TOF) stimulation, expressed as percentage of control first twitch, T1) during sevoflurane anesthesia for Caucasian participants.

DETAILED DESCRIPTION:
For most surgical procedures a depth of neuromuscular block of 1-2 twitches after TOF-stimulation is sufficient to avoid unwanted muscular activity. At reappearance of T2, the anesthesiologist might decide to either give (another) maintenance dose of rocuronium or vecuronium when surgery continues, to await spontaneous recovery of neuromuscular block or to reverse the neuromuscular block. Sugammadex has been shown in previous trials to greatly reduce the time to full recovery when administered at reappearance of T2, both after rocuronium- and vecuronium induced neuromuscular blockade. The current trial P05971 was conducted in Europe and set up to establish the dose response relationship of sugammadex given during sevoflurane anesthesia at reappearance of T2 after rocuronium or vecuronium in Caucasian participants. In addition to recovery time, also pharmacokinetics and safety of sugammadex were to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Is of American Society of Anesthesiologists (ASA) class 1 - 3;
* Is at least 20 years but under 65 years of age;
* Caucasian participants;
* Is scheduled for elective surgery requiring muscle relaxation in supine position and under sevoflurane anesthesia with an anticipated duration of about 1.5-3 hours;
* Has given written informed consent.

Exclusion criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Is known or suspected to have neuromuscular disorders impairing neuromuscular blocking (NMB) and/or significant renal dysfunction (for example a creatinine level > 1.6 mg/dl) and/or severe hepatic dysfunction.
* Is known or suspected to have a (family) history of malignant hyperthermia;
* Is known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Is receiving medication expected to interfere with the rocuronium or vecuronium given in this trial, based on the dose and time of administration;
* Females who were pregnant;
* Females of childbearing potential not using birth control or using only oral contraception as birth control;
* Was breast-feeding;
* Has already participated in P05971, or in another trial with sugammadex;
* Has participated in another clinical trial, not preapproved by the Sponsor, within 6 months of entering into P05971.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09-20 (Actual); Primary Completion 2006-08-31 (Actual); Study Completion 2006-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Puhringer FK, Gordon M, Demeyer I, Sparr HJ, Ingimarsson J, Klarin B, van Duijnhoven W, Heeringa M. Sugammadex rapidly reverses moderate rocuronium- or vecuronium-induced neuromuscular block during sevoflurane anaesthesia: a dose-response relationship. Br J Anaesth. 2010 Nov;105(5):610-9. doi: 10.1093/bja/aeq226. Epub 2010 Sep 28. PMID 20876699
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSr Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caucasian participants who had a surgical procedure using a general anesthesia of rocuronium or vecuronium for endotracheal intubation and maintenance of neuromuscular block were enrolled in this study.
Period: Overall Study
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Started | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Treated | 10 | 10 | 9 | 10 | 10 | 10 | 10 | 10 | 10 | 9
Completed | 10 | 10 | 9 | 9 | 10 | 8 | 10 | 10 | 8 | 9
Not Completed | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1
Not completed — Not Treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All Participants As Treated
Groups:
- Rocuronium + Placebo: After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
- Total: Total of all reporting groups
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex | Total
Number analyzed (Participants) | 10 | 10 | 9 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (7) | 52 (7) | 50 (9) | 49 (8) | 49 (13) | 48 (10) | 47 (9) | 46 (9) | 45 (10) | 47 (10) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 5 | 6 | 8 | 7 | 7 | 7 | 7 | 70
  Male | 2 | 2 | 2 | 5 | 4 | 2 | 3 | 3 | 3 | 2 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 9 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.9 (up to 24 hours)
Population: All randomized participants who received sugammadex or placebo; without any protocol violations, and who had at least one post baseline efficacy measurement, who had a TOF trace, had a reliable TOF trace, and where drug administration did not interfere with the effect of rocuronium or vecuronium.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 7 | 8 | 8 | 9 | 8 | 8 | 9 | 10 | 7 | 9
Minutes | 96.30 (33.13) | 16.30 (20.60) | 4.62 (5.97) | 1.43 (0.50) | 1.50 (0.40) | 79.02 (25.97) | 35.50 (42.13) | 5.07 (2.38) | 3.42 (1.85) | 3.03 (2.18)

2. Secondary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.7 (up to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 8 | 10 | 10 | 9 | 9
Minutes | 65.67 (35.73) | 3.08 (2.25) | 2.08 (1.12) | 1.12 (0.40) | 1.02 (0.12) | 58.12 (21.90) | 12.57 (24.48) | 2.35 (0.48) | 2.00 (1.25) | 1.70 (0.55)

3. Secondary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.8 (up to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 7 | 9 | 8 | 9 | 9 | 8 | 10 | 10 | 9 | 9
Minutes | 75.85 (36.65) | 6.25 (9.12) | 2.62 (1.80) | 1.28 (0.42) | 1.15 (0.25) | 64.33 (21.72) | 25.65 (35.40) | 3.10 (0.88) | 5.83 (11.43) | 2.12 (0.80)

ADVERSE EVENTS:
Time Frame: Up to 7 days after sugammadex or placebo treatment
Description: All randomized participants who received study treatment
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 1/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 1/10 | 0/10 | 0/10 | 2/10 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 6/9 | 10/10 | 10/10 | 8/10 | 10/10 | 6/10 | 9/10 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Placebo (N=10) | Rocuronium + 0.5 mg/kg Sugammadex (N=10) | Rocuronium + 1.0 mg/kg Sugammadex (N=9) | Rocuronium + 2.0 mg/kg Sugammadex (N=10) | Rocuronium + 4.0 mg/kg Sugammadex (N=10) | Vecuronium + Placebo (N=10) | Vecuronium + 0.5 mg/kg Sugammadex (N=10) | Vecuronium + 1.0 mg/kg Sugammadex (N=10) | Vecuronium + 2.0 mg/kg Sugammadex (N=10) | Vecuronium + 4.0 mg/kg Sugammadex (N=9)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Placebo (N=10) | Rocuronium + 0.5 mg/kg Sugammadex (N=10) | Rocuronium + 1.0 mg/kg Sugammadex (N=9) | Rocuronium + 2.0 mg/kg Sugammadex (N=10) | Rocuronium + 4.0 mg/kg Sugammadex (N=10) | Vecuronium + Placebo (N=10) | Vecuronium + 0.5 mg/kg Sugammadex (N=10) | Vecuronium + 1.0 mg/kg Sugammadex (N=10) | Vecuronium + 2.0 mg/kg Sugammadex (N=10) | Vecuronium + 4.0 mg/kg Sugammadex (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 3 (3) | 6 (7) | 4 (4) | 3 (3) | 4 (5) | 1 (1) | 2 (2) | 4 (4)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Postoperative constipation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 3 (3) | 6 (6) | 6 (7) | 4 (4) | 2 (2) | 3 (3) | 4 (6) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta 2 microglobulin urine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath holding (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital pruritus female (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning this clinical trial will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.